CLINICAL TRIAL: NCT04170985
Title: NeuroSeq: A Prospective Trial to Evaluate the Diagnostic Yield of Human Whole Genome Sequencing (WGS) Compared to Standard of Care in Adults With Suspected Genetic Neurological Disorders
Brief Title: NeuroSeq: A Prospective Trial to Evaluate the Diagnostic Yield of Whole Genome Sequencing (WGS) in Adult Neurology
Acronym: NeuroSEQ
Status: Completed | Type: Observational
Sponsor: Illumina, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Neuro-R001
Record Dates: First submitted 2019-11-18; First posted 2019-11-20 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Neurologic Deficits; Neurologic Disorder; Neurologic Abnormalities
MeSH Terms: conditions — Neurologic Manifestations; Nervous System Diseases; Nervous System Malformations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — EDTA tube will be collected for whole genome sequencing (WGS) testing and left-over de-identified samples will be retained for future research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single Cohort: All participants will receive cWGS testing revealed to the site PI/clinician at Day 180. Participants will all receive standard of care testing throughout the study.
  Interventions: Other: clinical Whole Genome Sequencing

INTERVENTIONS:
Other: clinical Whole Genome Sequencing — Participants will receive cWGS as well as standard of care testing. The clinician/site PI will be blinded to the cWGS results until Day 180.

SUMMARY:
Prospective, multi-site, single-arm study to evaluate the diagnostic yield of cWGS in adults with neurological disorders. A single cohort naive of genetic testing will receive standard of care testing for 180 days followed by cWGS. The cohort will be followed for a total of 365 days following enrollment.

DETAILED DESCRIPTION:
This is a prospective, randomized study to evaluate the diagnostic yield of SOC compared to cWGS in each participant. Throughout this study, each participant will receive SOC testing as determined by the site clinical team. After the physician orders SOC testing during standard clinical practice, the subject will be introduced and invited to participate in the study. On Day 180, the participant will receive a cWGS result and the participant will continue to be followed for an additional 180 days. A blood sample from each enrolled participant will be collected and shipped to the Illumina Clinical Services Laboratory ("ICSL"), which is Clinical Laboratory Improvement Amendments (CLIA)-certified and College of American Pathologists (CAP)-accredited. ICSL will conduct cWGS testing with the TruGenome Undiagnosed Disease Test ("TruGenome Test"). The TruGenome Test cWGS results will be provided to the Principal Investigator (PI) or designee who will evaluate each participant's test outcome based on aggregate medical information.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years at the time of consent
2. Participant is referred to a Neurogenetics Program due to suspected genetic etiology of a neurological syndrome
3. No history of prior genetic testing for the suspected condition in the participant or any family member with a similar phenotype
4. Must be able to have one - 4 to 6 ml tube of whole blood drawn for testing
5. Able to provide written consent. If participant unable to do so, a legally authorized representative (LAR) must do so on behalf of the participant

Exclusion Criteria:

1. Any known non-genetic cause(s) of disease, disorder, or phenotypic defect
2. Eligibility for enrollment of each participant is at the discretion of the site PI
3. Patient is unable or unwilling to undergo any form(s) of SOC genetic testing
4. SOC testing is NOT requested for the participant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A single cohort presenting with phenotypic symptoms of a suspected genetic neurological disorder who have been scheduled for Standard of Care (SOC) molecular testing as determined by their physician.
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2019-11-18 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Diagnostic Yield between cWGS and SOC testing | Day 0 - Day 365
  The number of participants who have a diagnosis in the SOC arm vs the cWGS arm as measured by the test outcome

SECONDARY OUTCOMES:
Change of Management between cWGS and SOC testing as measured by a management questionnaire collected on a case report form | Day 0 - Day 365
  The number of participants who have a change in management after receiving SOC results vs cWGS results as measured by a management questionnaire at baseline, Day 180 and Day 365
Resource Utilization between cWGS and SOC testing | Day 0 - Day 365
  The number of participants who have utilized resources to include specialist referrals, tests/procedures ordered and procedures avoided in the SOC arm vs the cWGS arm as measured by data collection case report forms
Quality of Life between cWGS and SOC testing | Day 0 - Day 365
  Comparison between Quality-of-Life scores as measured by the 12-Item Short Form Survey (SF12) from baseline compared to end of study
Diagnostic Accuracy between cWGS and SOC testing when comparing the medical monitor test outcome and the site PI test outcome | Day 0 - Day 180
  Diagnostic accuracy- percent positive agreement between test outcome classified by the medical monitor and the site PI or designee
Diagnostic Yield within Cohort when evaluating specific Neurologic disorders | Day 0 - Day 365
  Difference in diagnostic yield between cohorts of neurological disorders

OTHER OUTCOMES:
Time to Diagnosis between cWGS and SOC testing | Day 0 - Day 365
  Average time (in days) to diagnosis between SOC and cWGS testing (duration between when sample is approved and when result(s) is/are delivered)
Clinical Survey by the clinician who ordered SOC testing | Day 365
  Clinician and genetic counselor satisfaction measured by an end-of-study questionnaire determining the overall satisfaction with the use of cWGS testing
Participant Survey | Day 365
  Participant satisfaction measured by an end-of-study questionnaire determining the overall satisfaction with the use of cWGS testing Participant satisfaction measured by an end-of-study questionnaire determining the participant's overall satisfaction with the use of cWGS testing

CONTACTS AND LOCATIONS:
Overall Officials: Ryan J Taft, Ph.D, Study Chair — Illumina, Inc.
Locations (1):
- Univ. of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan in place to share data with other researchers.